CLINICAL TRIAL: NCT00904371
Title: Evaluation of the Effect of Telmisartan on Blood Pressure and Cardiovascular Risk Factor Index in High Risk Hypertensive Patients
Brief Title: Evaluation of the Effect of Telmisartan (Micardis® 80 mg/ MicardisPlus® 80/12.5 mg) on Blood Pressure and Cardiovascular Risk Factor Index in High Risk Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.585
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with arterial hypertention

SUMMARY:
The study is designed to evaluate the effect of treatment with Micardis/MicardisPlus on blood pressure and its ability to reduce different indicated cardiovascular risks. Further on, the study will evaluate the current antihypertensive treatment pattern in the daily practice among the patient population at increased cardiovascular risk.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of essential arterial hypertension (BP>140/90 mm HG or BP>130/80 mm Hg for diabetic patients)
* at least an additional cardiovascular risk factor

Exclusion criteria:

* hypersensitivity to the active substance or to any of the excipients in any ACE inhibitor or angiotensin receptor blocker (ARB) available on the local market
* pregnancy and lactation
* diseases involving biliary obstruction
* severe liver impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with arterial hypertension with moderate to very high cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- Slovenia (36):
  - Boehringer Ingelheim Investigational Site 24, Brežice
  - Boehringer Ingelheim Investigational Site 2, Brežice
  - Boehringer Ingelheim Investigational Site 12, Celje
  - Boehringer Ingelheim Investigational Site 16, Celje
  - Boehringer Ingelheim Investigational Site 17, Celje
  - Boehringer Ingelheim Investigational Site 1, Celje
  - Boehringer Ingelheim Investigational Site 33, Celje
  - Boehringer Ingelheim Investigational Site 18, Golnik
  - Boehringer Ingelheim Investigational Site 23, Golnik
  - Boehringer Ingelheim Investigational Site 29, Golnik
  - Boehringer Ingelheim Investigational Site 32, Golnik
  - Boehringer Ingelheim Investigational Site 15, Jesenice
  - Boehringer Ingelheim Investigational Site 4, Kranj
  - Boehringer Ingelheim Investigational Site 28, Litija
  - Boehringer Ingelheim Investigational Site 26, Ljubljana
  - Boehringer Ingelheim Investigational Site 35, Ljubljana
  - Boehringer Ingelheim Investigational Site 3, Ljubljana
  - Boehringer Ingelheim Investigational Site 6, Ljubljana
  - Boehringer Ingelheim Investigational Site 14, Maribor
  - Boehringer Ingelheim Investigational Site 22, Maribor
  - Boehringer Ingelheim Investigational Site 20, Murska Sobota
  - Boehringer Ingelheim Investigational Site 27, Murska Sobota
  - Boehringer Ingelheim Investigational Site 31, Murska Sobota
  - Boehringer Ingelheim Investigational Site 11, Novo Mesto
  - Boehringer Ingelheim Investigational Site 19, Novo Mesto
  - Boehringer Ingelheim Investigational Site 21, Novo Mesto
  - Boehringer Ingelheim Investigational Site 9, Novo Mesto
  - Boehringer Ingelheim Investigational Site 25, Sempeter
  - Boehringer Ingelheim Investigational Site 30, Sempeter
  - Boehringer Ingelheim Investigational Site 34, Sežana
  - Boehringer Ingelheim Investigational Site 10, Slovenj Gradec
  - Boehringer Ingelheim Investigational Site 36, Slovenj Gradec
  - Boehringer Ingelheim Investigational Site 13, Topolšica
  - Boehringer Ingelheim Investigational Site 5, Trbovlje
  - Boehringer Ingelheim Investigational Site 8, Trbovlje
  - Boehringer Ingelheim Investigational Site 7, Velenje

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase IV, Post Marketing Surveillance Study, non-interventional, multicentre, national, observational study in routine daily practice.
Period: Overall Study
Arm/Group | Micardis® 80mg; MicardisPlus® 80/12.5 mg
Started | 211
Completed | 202
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 4
Not completed — Discontinued at target blood pressure | 2
Not completed — Continued with Tritace | 1

BASELINE CHARACTERISTICS:
Arm/Group | Micardis® 80mg; MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 211
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.4)
Gender [Number; unit: Participants] — There were only 203 patients with non-missing gender
  Participants
    Female | 90
    Male | 113
Additional antihypertensive treatment at baseline [Number; unit: Percentage of participants] — Participants may have taken more than one antihypertensive treatment, so the percentages will not add to 100 percent.
  Percentage of participants
    ACE inhibitors | 19
    Diuretics | 15.2
    Calcium Channel Blockers | 26.5
    Beta Blockers | 39.3
    Other | 7.6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 204
mm Hg | -22.6 (17.1)

2. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 203
mm Hg | -10.1 (10.1)

3. Primary Outcome: Change From Baseline in SCORE (10 Year Risk for Fatal Cardiovascular Event)
Description: A 10 year risk of fatal cardiovascular disease (CVD) in populations at high risk. Minimum 0 percent risk to Maximum 47 percent risk.
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 172
units on a scale | -3.9 (8.8)

4. Primary Outcome: Change From Baseline in Framingham CVD Risk Assessment Score
Description: 10-year risk for hard coronary heart disease (CHD) outcomes (Myocardial Infarction and coronary death), according to Framingham Heart Study, measured in percent. Low risk (10 or less CHD risk at 10 years), intermediate risk (10-20), high risk (20 or more).
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 148
units on a scale | -7.6 (8.6)

5. Primary Outcome: Change From Baseline in Framingham Stroke Risk Assessment Score
Description: The risk assessment tool using data from the Framingham Heart Study to estimate 10-year risk for stroke, measured in percent. Low risk (10 or less stroke risk at 10 years), intermediate risk (10-20), high risk (20 or more).
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 146
units on a scale | -3.6 (8.0)

6. Primary Outcome: Change From Baseline in Risk Assessment According to ESH/ESC Guidelines
Description: ESH is the European society of hypertension, and ESC is the European society of cardiology.
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months)
Measure: Number; unit: Participants moved into category
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 139
Participants moved into category
  Average risk | 18
  Low added risk | 7
  Moderate added risk | -13
  Very high added risk | -12

7. Secondary Outcome: Pecentage of Patients That Achieved Target Blood Pressure (BP) Values According to ESH/ESC
Description: ESH/ESC a goal of treatment to be below values 130/80 mm/Hg for diabetic patients and below 140/90 mmHg for non-diabetic patients
Time Frame: 3rd visit (4-10 months)
Population: Patients with data at 3rd visit (4-10 months)
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 195
Percentage of participants
  Achieved target BP values | 32.8
  Not achieved target BP values | 67.2

8. Secondary Outcome: Additional Antihypertensive Treatment Pattern at Visit 3 (End of Study)
Description: Participants may have taken more than one antihypertensive treatment, so the percentages will not add to 100 percent.
Time Frame: 3rd visit (4-10 months)
Population: Patients with data at 3rd visit (4-10 months)
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 205
Percentage of participants
  ACE inhibitors | 19
  Diuretics | 11.2
  Calcium Channel Blockers | 32.2
  Beta Blockers | 36.1
  Other | 9.3

9. Secondary Outcome: Change in Heart Rate From Baseline to Study End
Time Frame: Baseline to 3rd visit (4-10 months)
Population: Patients with data both at baseline and on 3rd visit (4-10 months) and known diabetic status
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 156
Beats per minute | -3.2 (9.2)

10. Secondary Outcome: Number of Patients With Adverse Events (AE)
Time Frame: 4-10 months
Population: Treated patients
Measure: Number; unit: Participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 211
Participants | 4

11. Secondary Outcome: Number of Participants Not Completing Study
Description: Number of participants discontinuing study early for given reason
Time Frame: 3rd visit (4-10 months)
Population: Patients with data at 3rd visit (4-10 months)
Measure: Number; unit: Participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 211
Participants
  Adverse Event | 2
  Lost to follow up | 4
  Discontinued at target BP | 2
  Continued with Tritace | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Serious Adverse Events (participants affected / at risk) | 2/211
Other Adverse Events (participants affected / at risk) | 0/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micardis® 80mg MicardisPlus® 80/12.5 mg (N=211)
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip oedema (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.